CLINICAL TRIAL: NCT03611075
Title: Study to Evaluate and Explore Scales for Repetitive and Restricted Behaviors and Digital Biomarkers in Children, Adolescents, and Adults With Autism Spectrum Disorder (ASD)
Brief Title: A Study to Evaluate Scales for Repetitive and Restricted Behaviors in Children, Adolescents, and Adults With Autism Spectrum Disorder (ASD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BP40331; 2019-003524-20 (EudraCT Number)
Record Dates: First submitted 2018-07-11; First posted 2018-08-02 (Actual); Results first posted 2021-07-23 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Low-Functioning Autism Spectrum Disorder (ASD) Children (Experimental): Participants will be 5-12 years old, with Intelligence Quotient (IQ) scores between 50-70
  Interventions: Other: No Intervention
- High-Functioning ASD Children (Experimental): Participants will be 5-12 years old, with IQ scores of 70 or above
  Interventions: Other: No Intervention
- Low-Functioning ASD Adolescents (Experimental): Participants will be 13-17 years old, with IQ scores between 50-70
  Interventions: Other: No Intervention
- High-Functioning ASD Adolescents (Experimental): Participants will be 13-17 years old, with IQ scores of 70 or above
  Interventions: Other: No Intervention
- Low-Functioning ASD Adults (Experimental): Participants will be 18-45 years old, with IQ scores between 50-70
  Interventions: Other: No Intervention
- High-Functioning ASD Adults (Experimental): Participants will be 18-45 years old, with IQ scores of 70 or above
  Interventions: Other: No Intervention
- Typically Developing (TD) Healthy Participant Children (No Intervention): Participants will be 5-12 years old
- TD Healthy Participant Adolescents (No Intervention): Participants will be 13-17 years old
- TD Healthy Participant Adults (No Intervention): Participants will be 18-45 years old

INTERVENTIONS:
Other: No Intervention — No interventions are administered in this study
  Arms: High-Functioning ASD Adolescents; High-Functioning ASD Adults; High-Functioning ASD Children; Low-Functioning ASD Adolescents; Low-Functioning ASD Adults; Low-Functioning Autism Spectrum Disorder (ASD) Children

SUMMARY:
This is a non-drug study seeking to characterize different scales to measure repetitive and restrictive behaviors in different ASD sub-populations over time. This study will also explore the use of digital biomarkers.

ELIGIBILITY:
Inclusion Criteria for All Participants

* Males and females
* Availability of a parent or other reliable caregiver. The same person must agree to accompany the participant to all clinic visits and provide information about the participant's behavior and symptoms

Inclusion Criteria for Participants with Autism Spectrum Disorders (ASD)(Diagnostic evaluations will be completed at study site by research staff and supervised by a licensed psychologist)

* Age: 5-45 years
* Diagnosis of ASD based on the Diagnostic and Statistical Manual of Mental Disorders (DSM-5), and the Autism Diagnostic Observation Schedule (ADOS-2).
* Children's Yale-Brown Obsessive Compulsive Scale modified for ASD (CY-BOCS-ASD) total score of at least 12
* Clinical Global Impression-Severity (CGI-S) scale of at least 4 about participant's current autism severity
* Intelligence quotient (IQ) score of 50 or above as assessed by the Abbreviated Intelligence Quotient (ABIQ) SB5 scale
* All medications and treatments are expected to be stable for the duration of the study

Inclusion Criteria for Typically Developing (TD) Healthy Participants

-TD participants aged 5-45 years

Exclusion Criteria for All Participants

* Participation in an in investigational drug or device study within 4 weeks or 5 times the half-life of the investigational molecule prior to screening, and participant is not expected to enroll in any other trial during the study
* Co-occurring disease, condition, or treatment that might interfere with the conduct of the study or pose an unacceptable risk to the participant
* Unstable or uncontrolled clinically significant psychiatric and/or neurological disorder that may interfere with study objectives

Exclusion Criteria for Participants with ASD -Known "syndromic" ASD (e.g. Fragile X syndrome, Angelman syndrome, Prader-Willi, Rett's syndrome, tuberous sclerosis, Dup15q syndrome) History of alcohol misuse and/or illicit drug use during the last 12 months of the study

Exclusion Criteria for TD Healthy Participants

-TD healthy participants with a first-degree relative with ASD

Ages: 5 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 144 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2020-05-21 (Actual); Study Completion 2020-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (18):
- United States (15):
  - Harmonex Neuroscience Research, Dothan, Alabama
  - Southwest Autism Research and Resource Center, Phoenix, Arizona
  - PCSD Feighner Research, San Diego, California
  - Stanford University School of Medicine, Stanford, California
  - Clinical Neuroscience Solutions Inc; Jacksonville Clinic, Jacksonville, Florida
  - University of Minnesota; Clin. Neuro Research Unit, Minneapolis, Minnesota
  - Nathan S. Kline Institute for Psychiatric Research, Orangeburg, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - BioBehavioral Research of Austin, PC, Austin, Texas
  - Red Oak Psychiatry Associates, PA, Houston, Texas
  - Road Runner Research Ltd, San Antonio, Texas
  - Northwest Clinical Research Center - ClinEdge - PPDS, Bellevue, Washington
  - Seattle Children's Hospital - PIN; Investigational Drug Services, Seattle, Washington
- Holland Bloorview Kids Rehabilitation Hospital; Autism Research Centre, East York, Ontario, Canada
- United Kingdom (2):
  - Gartnavel Royal Hospital; Mental Health & Wellbeing, Glasgow
  - Kings College London, London

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 227 participants were screened, of these, 83 participants were screen failures
Pre-assignment Details: A total of 144 participants were enrolled at 18 centers in the following countries: United States (15 sites), United Kingdom (2 sites), and Canada (1 site). The 144 participants included 95 participants with Autism Spectrum Disorder (ASD) and 49 Typically Developing (TD) healthy participants.
Groups:
- High-Functioning Autism Spectrum Disorder (ASD) Children; Healthy Control Participants Children: Participants will be 5-12 years old, with IQ scores of 70 or above
- Healthy Control Participants Adolescents: Participants will be 13-17 years old, with IQ scores of 70 or above
- Healthy Control Participants Adults: Participants will be 18-45 years old, with IQ scores of 70 or above
Period: Overall Study
Arm/Group | High-Functioning Autism Spectrum Disorder (ASD) Children | High-Functioning ASD Adolescents | High-Functioning ASD Adults | Low-Functioning Autism Spectrum Disorder (ASD) Children | Low-Functioning ASD Adolescents | Low-Functioning ASD Adults | Healthy Control Participants Children | Healthy Control Participants Adolescents | Healthy Control Participants Adults
Started | 16 | 15 | 16 | 17 | 13 | 18 | 15 | 17 | 17
Completed | 15 | 13 | 14 | 13 | 13 | 18 | 13 | 17 | 17
Not Completed | 1 | 2 | 2 | 4 | 0 | 0 | 2 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Reason unknown | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- High-Functioning ASD Children: Participants will be 5-12 years old, with Intelligence Quotient (IQ) scores between 50-70
- Healthy Control Participants Adolescence: Participants will be 13-17 years old, with IQ scores of 70 or above
- Healthy Control Participants Adults: High-Functioning ASD AdultsEdit Participants will be 18-45 years old, with IQ scores of 70 or above
- Total: Total of all reporting groups
Arm/Group | Low-Functioning Autism Spectrum Disorder (ASD) Children | Low-Functioning ASD Adolescents | Low-Functioning ASD Adults | High-Functioning ASD Children | High-Functioning ASD Adolescents | High-Functioning ASD Adults | Healthy Control Participants Children | Healthy Control Participants Adolescence | Healthy Control Participants Adults | Total
Number analyzed (Participants) | 17 | 13 | 18 | 16 | 15 | 16 | 15 | 17 | 17 | 144
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.6 (1.9) | 15.2 (1.4) | 15.2 (1.4) | 9.6 (2.3) | 15.1 (1.4) | 24.6 (6.0) | 8.5 (2.1) | 14.8 (1.4) | 31.2 (7.0) | 17.1 (8.7)
Sex/Gender, Customized [Number; unit: Participants]
  Male | 14 | 12 | 14 | 14 | 12 | 12 | 6 | 10 | 2 | 96
  Female | 3 | 1 | 4 | 2 | 3 | 4 | 9 | 7 | 15 | 48
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 7 | 5 | 2 | 4 | 3 | 2 | 4 | 2 | 4 | 33
  Not Hispanic or Latino | 10 | 8 | 15 | 12 | 11 | 14 | 11 | 14 | 13 | 108
  Unknown | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
  Not stated | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  Black or African American | 4 | 3 | 1 | 7 | 1 | 0 | 3 | 1 | 3 | 23
  White | 13 | 8 | 16 | 9 | 11 | 14 | 11 | 12 | 12 | 106
  Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
  Asian | 0 | 2 | 1 | 0 | 1 | 2 | 0 | 3 | 2 | 11
  Multiple | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Children's Yale-Brown Obsessive Compulsive Scale Modified for Autism Spectrum Disorder (CY-BOCS-ASD) - Total Score
Description: The CY-BOCS-ASD is where the interviewer asks the parent/caregiver about past and present repetitive behaviors, guided by the revised repetitive behavior checklist with a list of 25 behaviors, classified into the following categories: Hoarding/ritualistic behavior, Sensorymotor and arranging, Insistence on routines /Self-injurious behaviors, Stereotypy and Restricted interests. This checklist was expanded to include repetitive behaviors commonly seen in children with ASD. A target symptom list comprising the four most troublesome behaviors is established by the interviewer. The severity (0 to 4) of each target behavior is rated for the following five items: time spent, interference, distress, resistance and degree of control to generate a total score (0-20). The ratings evaluate the symptom severity over the past week and are based on the information collected from the child and parent/caregiver during the interview. Values at visits are reported.
Time Frame: Baseline, Weeks 2 and 12
Population: Autism Spectrum Disorder (ASD) Population
Measure: Mean (Standard Deviation); unit: Score on a Scale
Groups:
- Low-Functioning ASD Children: Participants will be 5-12 years old, with Intelligence Quotient (IQ) scores between 50-70
Arm/Group | High-Functioning ASD Children | High-Functioning ASD Adolescents | High-Functioning ASD Adults | Low-Functioning ASD Children | Low-Functioning ASD Adolescents | Low-Functioning ASD Adults
Number analyzed (Participants) | 16 | 15 | 16 | 17 | 13 | 18
Score on a Scale
  Baseline | 14.81 (2.40) | 14.60 (2.77) | 14.94 (1.95) | 15.71 (1.61) | 15.23 (2.24) | 15.83 (2.12)
  Week 2: number analyzed (Participants) | 16 | 13 | 15 | 13 | 12 | 18
  Week 2 | 15.06 (2.89) | 13.69 (2.93) | 13.00 (3.36) | 15.15 (2.30) | 14.67 (4.44) | 15.50 (2.36)
  Week 12: number analyzed (Participants) | 15 | 13 | 14 | 12 | 13 | 18
  Week 12 | 15.13 (3.09) | 12.77 (3.77) | 13.36 (2.59) | 15.58 (1.68) | 14.00 (3.37) | 14.44 (2.81)

2. Primary Outcome: Montefiore Einstein Rigidity Scale (MERS-R)
Description: The MERS-R was to assess 3 domains of rigid behavior in children and adults. It's a clinician-administered scale in which the clinician uses all available information to rate. Each domains is assessed separately, during examples are discussed and related behaviors are probed for more individualized exemplars. A list of relevant behaviors is compiled for each domain, and ratings for the items are based on the average occurrence of the behaviors over the past one week. Total values at visits are reported and domains are assessed: ASD: 1. Behavioral Rigidity (e.g., insistence on sameness, things must be done in his/her way) 2. Cognitive Rigidity (e.g., inflexible adherence to rules) 3. Protest (in response to deviation from rigidity; e.g., verbal objection, tantrum, physical aggression). These domain scores can range from 0 (no problems) to 4 (severe problems). The total score represents the sum of the domain scores ranging from 0-48, where higher scores indicate more severe problems.
Time Frame: Baseline, Weeks 2 and 12
Population: ASD Population. "Number of Participants Analyzed" is the total number of participants enrolled at baseline, "Number Analyzed" is number of participants evaluable.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | High-Functioning ASD Children | High-Functioning ASD Adolescents | High-Functioning ASD Adults | Low-Functioning ASD Children | Low-Functioning ASD Adolescents | Low-Functioning ASD Adults
Number analyzed (Participants) | 16 | 15 | 16 | 17 | 13 | 18
Score on a Scale
  Baseline | 29.88 (8.30) | 25.67 (7.09) | 22.56 (7.83) | 28.35 (7.13) | 25.46 (7.81) | 25.78 (6.92)
  Week 2: number analyzed (Participants) | 16 | 13 | 15 | 14 | 12 | 18
  Week 2 | 28.81 (7.32) | 22.77 (8.93) | 21.07 (8.28) | 27.86 (6.85) | 26.83 (10.30) | 26.67 (7.81)
  Week 12: number analyzed (Participants) | 15 | 13 | 14 | 13 | 13 | 18
  Week 12 | 27.87 (8.63) | 21.15 (8.82) | 20.64 (7.04) | 25.69 (4.97) | 24.08 (9.54) | 24.67 (8.53)

3. Primary Outcome: Repetitive Behavior Scale-Revised (RBS-R)
Description: The Repetitive Behavior Scale-Revised (RBS-R) is a 43-item caregiver-report questionnaire to measure breadth of repetitive behaviors in children, adolescents, and adults with ASD. It provides a quantitative measure of the full spectrum of repetitive behaviors of 6 subscales: Stereotype, Self-injurious, Compulsive, Ritualistic, Sameness and Restricted Behaviors. Caregivers are asked to read a list of behaviors and choose for each item a score that best describes how much of a problem the behavior has been over the last month. Behaviors are rated on a 4-point scale: 0-Behavior does not occur, 1-Behavior occurs and is a mild problem, 2-Behavior occurs and is a moderate problem, 3-Behavior occurs and is a severe problem. The total score is the sum of all 43 items and can range from 0 to 129. Higher scores indicate more severe problems with repetitive behaviors. The sums of score values at visits are reported.
Time Frame: Baseline, Weeks 2 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | High-Functioning ASD Children | High-Functioning ASD Adolescents | High-Functioning ASD Adults | Low-Functioning ASD Children | Low-Functioning ASD Adolescents | Low-Functioning ASD Adults
Number analyzed (Participants) | 16 | 15 | 16 | 17 | 13 | 18
Score on a Scale
  Baseline: number analyzed (Participants) | 16 | 14 | 16 | 17 | 12 | 18
  Baseline | 39.81 (21.00) | 38.29 (19.77) | 33.06 (19.39) | 56.82 (25.62) | 38.25 (21.82) | 42.67 (22.89)
  Week 2: number analyzed (Participants) | 16 | 13 | 15 | 14 | 11 | 18
  Week 2 | 40.88 (22.51) | 37.31 (18.00) | 32.27 (21.10) | 54.00 (27.17) | 38.18 (25.23) | 40.17 (24.86)
  Week 12: number analyzed (Participants) | 15 | 12 | 14 | 13 | 12 | 18
  Week 12 | 36.07 (21.24) | 36.25 (18.24) | 33.07 (20.99) | 51.00 (24.70) | 36.33 (21.96) | 37.78 (23.09)

4. Primary Outcome: Repetitive Behavior Questionnaire for Children (RBQ-2)
Description: The RBQ-2 is a 20 items questionnaire to assess the spectrum of restricted and repetitive behaviors observed in individuals with ASD such as repetitive motor movements, rigidity/adherence to routine, preoccupation with restricted patterns of interest and unusual sensory Interest (Leekman et al 2007; Honey et al 2012). The RBQ-2 exists in two different versions, a caregiver reported version for pediatric subjects RBQ-2 and a participant-reported version for adults RBQ-2A (Barrett et al 2015). The RBQ-2, the caregiver version is used for this reported data set. To ensure for this study a comparable the mean total score is calculated as the sum of the items, total scores at visits are reported. For the RBQ-2, the possible total score can range between 20-60, with higher scores indicating more frequent RRB.
Time Frame: Baseline, Weeks 2 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | High-Functioning ASD Children | High-Functioning ASD Adolescents | High-Functioning ASD Adults | Low-Functioning ASD Children | Low-Functioning ASD Adolescents | Low-Functioning ASD Adults
Number analyzed (Participants) | 16 | 15 | 16 | 17 | 13 | 18
Score on a Scale
  Baseline: number analyzed (Participants) | 16 | 14 | 10 | 17 | 12 | 14
  Baseline | 38.63 (8.16) | 35.57 (8.61) | 34.50 (8.45) | 41.76 (9.03) | 38.00 (8.54) | 39.14 (7.68)
  Week 2: number analyzed (Participants) | 16 | 13 | 10 | 14 | 11 | 17
  Week 2 | 38.00 (8.10) | 37.62 (8.17) | 35.80 (4.32) | 41.86 (8.84) | 39.36 (8.82) | 37.12 (6.86)
  Week 12: number analyzed (Participants) | 15 | 12 | 10 | 13 | 12 | 15
  Week 12 | 35.80 (8.15) | 36.42 (7.88) | 35.10 (7.62) | 43.00 (8.77) | 37.17 (8.35) | 38.20 (8.37)

5. Primary Outcome: Restricted Behavior Questionnaire for Adults (RBQ-2A)
Description: The RBQ-2 is a 20 items questionnaire to assess the spectrum of restricted and repetitive behaviorsobserved in individuals with ASD such as repetitive motor movements, rigidity/adherence to routine, preoccupation with restricted patterns of interest and unusual sensory Interest (Leekman et al 2007; Honey et al 2012). The RBQ-2 exists in two different versions, a caregiver reported version for pediatric subjects RBQ-2 and a participant-reported version for adults RBQ-2A (Barrett et al 2015). The RBQ-2, the caregiver version is used for this reported data set. Total score is calculated as the sum of the items, total scores at visits are reported. For the RBQ-2A, the possible total score can range between 20 to 60, with higher scores indicating more frequent and severe RRB.
Time Frame: Baseline, Weeks 2 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | High-Functioning ASD Adolescents | High-Functioning ASD Adults | Low-Functioning ASD Adolescents | Low-Functioning ASD Adults
Number analyzed (Participants) | 15 | 16 | 13 | 18
Score on a Scale
  Baseline: number analyzed (Participants) | 14 | 14 | 2 | 15
  Baseline | 36.29 (6.07) | 39.00 (11.18) | 35.50 (9.19) | 40.73 (6.93)
  Week 2: number analyzed (Participants) | 12 | 14 | 1 | 15
  Week 2 | 38.25 (6.15) | 41.86 (10.34) | 43.00 (0) | 39.60 (8.64)
  Week 12: number analyzed (Participants) | 12 | 13 | 3 | 16
  Week 12 | 37.67 (5.18) | 41.54 (11.03) | 36.33 (7.09) | 42.00 (7.47)

6. Primary Outcome: Childhood Routines Inventory-Revised (CRI-R)
Description: The CRI-R (for children and adolescents) and ARI (for adults) were developed together and are closely related scales (Evans et al 2017).The CRI-R and ARI questionnaires capture a wide range of restricted and repetitive behaviors, including stereotypies, tics, compulsions, habits, sensory sensitivities, and focused interests, in the context of typical and atypical development in children, adolescents and adults across the entire lifespan. All items will be answered on a five-point Likert scale from not at all/ never, a little/rarely, somewhat/ sometimes, quite a lot/ often, and very much / always. The caregiver-completed CRI-R scale for pediatric subjects includes 62 items. Total score is calculated as the sum of the items, total scores at visits are reported.
  For the CRI-R, the possible total score can range between 62 - 310, with higher scores indicating more frequent RRB.
Time Frame: Baseline, Weeks 2 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | High-Functioning ASD Children | High-Functioning ASD Adolescents | High-Functioning ASD Adults | Low-Functioning ASD Children | Low-Functioning ASD Adolescents | Low-Functioning ASD Adults
Number analyzed (Participants) | 16 | 15 | 16 | 17 | 13 | 18
Score on a Scale
  Baseline: number analyzed (Participants) | 16 | 14 | 8 | 16 | 12 | 14
  Baseline | 177.38 (35.05) | 174.50 (49.25) | 166.25 (44.84) | 187.69 (40.81) | 164.33 (40.58) | 171.21 (40.16)
  Week 2: number analyzed (Participants) | 16 | 13 | 9 | 14 | 11 | 16
  Week 2 | 172.44 (35.78) | 173.62 (48.74) | 165.00 (40.68) | 189.93 (44.06) | 161.09 (37.42) | 170.38 (36.86)
  Week 12: number analyzed (Participants) | 16 | 12 | 9 | 13 | 12 | 14
  Week 12 | 170.27 (45.35) | 168.42 (51.16) | 162.22 (48.66) | 185.69 (39.90) | 155.08 (37.46) | 171.50 (39.60)

7. Primary Outcome: Adult Routines Inventory (ARI)
Description: The CRI-R (for children and Adolescents) and ARI (for adults) were developed together and are closely related scales (Evans et al 2017).The CRI-R and ARI questionnaires capture a wide range of RRBs, including stereotypies, tics, compulsions, habits, sensory sensitivities, and focused interests, in the context of typical and atypical development in children, adolescents and adults across the entire lifespan. All items will be answered on a five-point Likert scale from not at all/ never, a little/rarely, somewhat/ sometimes, quite a lot/ often, and very much / always. The caregiver-completed CRI-R scale for pediatric subjects includes 62 items. The participant-reported ARI scale for adult subjects includes 55 items and will be completed by the participant. Total score is calculated as the sum of the items, mean total scores at visits are reported.
  For the ARI, the possible total score can range between 55-275, with higher scores indicating more frequent RRB.
Time Frame: Baseline, Weeks 2 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | High-Functioning ASD Adolescents | High-Functioning ASD Adults | Low-Functioning ASD Adolescents | Low-Functioning ASD Adults
Number analyzed (Participants) | 15 | 16 | 13 | 18
Score on a Scale
  Baseline: number analyzed (Participants) | 14 | 15 | 1 | 15
  Baseline | 142.50 (31.00) | 166.00 (40.85) | 165.00 (0) | 158.07 (22.41)
  Week 2: number analyzed (Participants) | 12 | 14 | 1 | 15
  Week 2 | 137.00 (28.90) | 164.00 (43.35) | 165.00 (0) | 150.40 (22.47)
  Week 12: number analyzed (Participants) | 12 | 13 | 3 | 16
  Week 12 | 140.67 (34.25) | 159.15 (46.74) | 144.33 (10.69) | 155.56 (27.97)

8. Secondary Outcome: Clinical Global Impression Scales (CGI)
Description: The CGI rating scales are tools used to evaluate both the severity of illness and change from Baseline (Guy et al 1976). The CGI-S reflects the rater's impression of the participant's current autism severity on a 7-point scale ranging from no symptoms (1) to very severe symptoms (7). The CGI-I is used to assess the clinical change as compared to symptoms at Baseline using a 7-point scale, ranging from very much improved (1) to very much worse (7). For this study modified versions will be used (Busner et al 2007 and 1991; Busner et al 1997). Values at visits are reported.
Time Frame: Baseline, Weeks 2 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | High-Functioning ASD Children | High-Functioning ASD Adolescents | High-Functioning ASD Adults | Low-Functioning ASD Children | Low-Functioning ASD Adolescents | Low-Functioning ASD Adults
Number analyzed (Participants) | 16 | 15 | 16 | 17 | 13 | 18
Score on a Scale
  Baseline | 4.63 (0.50) | 4.47 (0.83) | 4.56 (0.73) | 5.18 (0.73) | 5.69 (0.75) | 4.89 (0.76)
  Week 2: number analyzed (Participants) | 16 | 13 | 15 | 14 | 12 | 18
  Week 2 | 4.63 (0.62) | 4.46 (0.78) | 4.60 (0.74) | 5.14 (0.86) | 5.58 (0.90) | 4.94 (0.73)
  Week 12: number analyzed (Participants) | 15 | 13 | 14 | 13 | 13 | 17
  Week 12 | 4.73 (0.59) | 4.38 (0.65) | 4.64 (0.74) | 5.08 (0.86) | 5.46 (0.88) | 4.82 (0.81)

9. Secondary Outcome: Child's Sleep Habits Questionnaire (CSHQ)
Description: The CSHQ is a 54-item parent or caregiver-reported measure that enquires about children's sleep habits and possible difficulties with sleep (Owens et al 2000). A subsequent study supported the validity of the CSHQ in children as young as 2 years. Using a 3-point Likert scale parents indicate whether a behavior occurs usually = 3, (i.e. 5 or more times a week),sometimes = 2 (i.e. 2-4 times a week) or rarely = 1 (i.e. 0-1 times a week). The summation of the frequency rating creates the total score, with higher scores reflecting greater sleep disturbances. The total score is calculated as the sum of a subset of 33 items and can range from 33 - 99, with higher scores reflecting greater sleep disturbances. Total scores at each visit are reported.
Time Frame: Baseline, Weeks 2 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a Sclae
Arm/Group | High-Functioning ASD Children | High-Functioning ASD Adolescents | High-Functioning ASD Adults | Low-Functioning ASD Children | Low-Functioning ASD Adolescents | Low-Functioning ASD Adults
Number analyzed (Participants) | 16 | 15 | 18 | 17 | 13 | 16
Score on a Sclae
  Baseline: number analyzed (Participants) | 16 | 13 | 11 | 16 | 11 | 6
  Baseline | 54.00 (8.18) | 48.08 (10.05) | 42.73 (7.32) | 48.31 (9.56) | 41.45 (3.80) | 40.33 (4.89)
  Week 2: number analyzed (Participants) | 16 | 13 | 15 | 14 | 10 | 8
  Week 2 | 54.19 (6.42) | 50.00 (9.69) | 43.40 (6.42) | 47.07 (10.59) | 42.90 (3.51) | 40.50 (2.98)
  Week 12: number analyzed (Participants) | 15 | 12 | 14 | 13 | 12 | 8
  Week 12 | 53.87 (8.11) | 47.58 (9.35) | 43.79 (8.79) | 45.23 (7.43) | 41.58 (3.60) | 39.25 (5.23)

10. Secondary Outcome: Pittsburg Sleep Quality Index (PSQI)
Description: The PSQI assesses sleep quality during the previous month (Buysse et al 1989). It consists of 19 self-rated questions. A wide variety of factors relating to sleep quality are assessed, including estimates of sleep duration and latency and the frequency and severity of specific sleep-related problems. These 19 items are grouped into seven component scores, each weighted equally on a 0-3 scale. The global PSQI score has a range of 0-21 and higher scores indicate worse sleep quality. Adult participants with a mental age of at least 10 years and adolescents deemed able to complete the PSQI will complete this scale.
Time Frame: Baseline, Weeks 2 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | High-Functioning ASD Adolescents | High-Functioning ASD Adults | Low-Functioning ASD Adolescents | Low-Functioning ASD Adults
Number analyzed (Participants) | 15 | 16 | 13 | 18
Score on a Scale
  Baseline: number analyzed (Participants) | 14 | 15 | 1 | 13
  Baseline | 6.00 (3.33) | 7.67 (3.79) | 2.00 (0) | 6.69 (2.95)
  Week 2: number analyzed (Participants) | 12 | 15 | 1 | 15
  Week 2 | 6.33 (3.75) | 6.60 (3.64) | 6.00 (0) | 6.40 (3.00)
  Week 12: number analyzed (Participants) | 12 | 13 | 3 | 16
  Week 12 | 5.75 (4.45) | 7.15 (3.58) | 5.67 (3.51) | 4.88 (3.46)

11. Secondary Outcome: Reading the Mind in the Eyes Test -R (RMET-R)
Description: RMET was used as anchor for the analysis of digital biomarker data and therefore also healthy participants should complete the RMET. However, at study start, it will be decided for each individual participant if the RMET-R or RMET-C should be used or if neither of the two RMET versions is deemed appropriate for the participant.
  In RMET-R, the participants are presented a series of 36 pictures of the eye-region of the face of different individuals, and are asked to choose which of four words best describes what the person in the photograph is thinking or feeling. This test was conceived of as a test of how well the participant can put themselves into the mind of the other person, and "tune in" to their mental state. The sum of the correct answers at each visit are reported as the total score. The total score can range from 0-36, and the higher the score, the more the participant can put themselves into the mind of the other person etc.
Time Frame: Baseline, Week 12
Population: High functioning adolescents and adults as well as low functioning adult ASD Population participated. Not all participants were available at baseline and Week 12 timepoints. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | High-Functioning ASD Adolescents | High-Functioning ASD Adults | Low-Functioning ASD Adults
Number analyzed (Participants) | 15 | 16 | 18
Score on a Scale
  Baseline: number analyzed (Participants) | 9 | 11 | 9
  Baseline | 15.44 (2.88) | 21.45 (8.37) | 12.00 (4.95)
  Week 12: number analyzed (Participants) | 8 | 9 | 9
  Week 12 | 15.63 (4.53) | 19.22 (8.89) | 10.67 (4.39)

12. Secondary Outcome: Reading the Mind in the Eyes Test Child -C (RMET-C)
Description: RMET was used as anchor data for analysis of digital biomarkers and therefore also healthy participants should complete the RMET. However at study start it will be decided for each individual participant if the RMET-R or RMET-C should be used or if neither of the two RMET versions is deemed appropriate for the participant.
  In the shorter pediatric RMET-C, the participants are presented a series of 28 pictures of the eye-region of the face of different individuals, and are asked to choose which of four words best describes what the person in the photograph is thinking or feeling. This test was conceived of as a test of how well the participant can put themselves into the mind of the other person, and "tune in" to their mental state. The sum of the correct answers at each visit is reported as total scores.
  For the RMET-C the total score can range from 0-28, and the higher the score, the more the participant can put themselves into the mind of the other person etc.
Time Frame: Baseline, Week 12
Population: ASD Population participated. Not all participants were available at baseline and Week 12 timepoints. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | High-Functioning ASD Children | High-Functioning ASD Adolescents | High-Functioning ASD Adults | Low-Functioning Autism Spectrum Disorder (ASD) Children | Low-Functioning ASD Adolescents | Low-Functioning ASD Adults
Number analyzed (Participants) | 16 | 15 | 16 | 17 | 13 | 18
Score on a Scale
  Baseline: number analyzed (Participants) | 11 | 12 | 3 | 9 | 6 | 5
  Baseline | 16.64 (5.26) | 16.25 (3.22) | 12.67 (5.69) | 11.00 (3.46) | 14.33 (3.93) | 15.00 (5.83)
  Week 12: number analyzed (Participants) | 12 | 9 | 4 | 8 | 5 | 4
  Week 12 | 17.33 (6.57) | 15.78 (4.15) | 14.00 (4.00) | 10.63 (4.00) | 11.40 (5.41) | 14.75 (6.08)

13. Secondary Outcome: Hamilton Anxiety Rating Scale (HAM-A)
Description: The HAM-A is a clinician-rated scale to analyze the severity of symptoms of anxiety. The HAM-A consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). The scale is intended for adults, adolescents, and children´(Hamilton et al 1959). The HAM-A will be completed only for adult participants in this study.
  Each of the 14 items is scored on a scale of 0 (not present) to 4. (severe) The total score is calculated as the sum of all items. The total score can range from 0-56, where <17 indicates mild severity, 18-24 mild to moderate, ≥ 24 severe anxiety. The total scores at each visit are reported (scores ≤ 7 were considered to represent no/minimal).
Time Frame: Baseline, Weeks 2 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | High-Functioning ASD Adults | Low-Functioning ASD Adults
Number analyzed (Participants) | 16 | 18
Score on a Scale
  Baseline: number analyzed (Participants) | 16 | 16
  Baseline | 10.81 (6.64) | 11.00 (9.32)
  Week 2: number analyzed (Participants) | 12 | 16
  Week 2 | 11.46 (7.80) | 7.19 (4.82)
  Week 12: number analyzed (Participants) | 12 | 16
  Week 12 | 9.92 (7.56) | 6.25 (5.84)

14. Secondary Outcome: Parent Rated Anxiety Scale for ASD (PRAS-ASD)
Description: PRAS-ASD is a caregiver-rated scale with 25 items to assess the severity of anxiety symptoms in children and adolescents with ASD. Caregivers are asked to describe their child's worries and anxiety-related behaviors over the past two weeks on a 0 to 3-point scale from NONE=not present; MILD=Present sometimes, not a real problem; MODERATE=Often present and a problem; SEVERE=Very frequent and a major problem. A publication about the PRAS-ASD is in preparation (as per personal communication, Prof Dr. Lawrence Scahill at Emory University). The PRAS-ASD will be completed for children and adolescents. Each of the 25 items is scored by the caregiver on a scale of 0 (None) to 3. (severe) The total score is calculated as the sum of all items. The total score can range from 0-75. , where higher scores indicate more severe anxiety. The total scores at each visit are reported.
Time Frame: Baseline, Weeks 2 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | High-Functioning ASD Children | High-Functioning ASD Adolescents | Low-Functioning ASD Children | Low-Functioning ASD Adolescents
Number analyzed (Participants) | 16 | 15 | 17 | 13
Score on a Scale
  Baseline: number analyzed (Participants) | 16 | 14 | 12 | 12
  Baseline | 33.94 (18.03) | 28.50 (17.33) | 29.12 (17.80) | 21.92 (13.97)
  Week 2: number analyzed (Participants) | 16 | 13 | 14 | 11
  Week 2 | 29.38 (17.69) | 29.15 (17.64) | 28.79 (17.30) | 21.36 (13.48)
  Week 12: number analyzed (Participants) | 15 | 11 | 13 | 11
  Week 12 | 28.53 (16.50) | 25.91 (20.29) | 25.46 (15.90) | 21.18 (13.00)

15. Secondary Outcome: Beck Anxiety Index (BAI)
Description: The Beck Anxiety Inventory (BAI) consists of 21 self-reported items (four-point scale) used to assess the intensity of physical and cognitive anxiety symptoms during the past week. Scores may range from 0 to 63: minimal anxiety levels (0-7), mild anxiety (8-15), moderate anxiety (16-25), and severe anxiety (26-63). Each item contains four possible responses, which range in severity from 0=not at all to 3=severely, I could barely stand it. Participants are asked to provide answers based on the way they have been feeling over the past month, including the assessment day. Adult participants were asked to complete the BAI. Adolescent participants completed the BAI if deemed appropriate by Investigator for the individual participant based on mental age. The BAI is a self-administered scale and the sum values at visits are reported as total scores. The total score can range from 0-63. The higher score values indicate more anxiety symptoms.
Time Frame: Baseline, Weeks 2 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | High-Functioning ASD Adolescents | High-Functioning ASD Adults | Low-Functioning ASD Adolescents | Low-Functioning ASD Adults
Number analyzed (Participants) | 15 | 16 | 13 | 18
Score on a Scale
  Baselin: number analyzed (Participants) | 13 | 14 | 1 | 15
  Baselin | 17.21 (12.41) | 19.64 (12.32) | 16.00 (0) | 13.47 (10.56)
  Week 2: number analyzed (Participants) | 12 | 14 | 1 | 15
  Week 2 | 12.08 (9.43) | 15.50 (14.65) | 16.00 (0) | 16.53 (11.88)
  Week 12: number analyzed (Participants) | 12 | 13 | 3 | 16
  Week 12 | 13.33 (7.55) | 16.92 (14.78) | 8.33 (2.52) | 14.94 (10.68)

16. Secondary Outcome: Digital Biomarkers
Description: It's to measure behaviors and symptoms related to ASD remotely with digital biomarkers, based on adherence (number of participants adhered) to the digital biomarker schedule of assessments. Participants will use a dedicated smartphone and wearable device to perform at-home exploratory measures in Digital Biomarker Adherence measurement. It consisted of surveys and performance outcome measures related to autism-associated symptoms, as well as continuous passive monitoring of participant behavior. Percentage of participants adhered were reported per assessment including Active Test, Conversation, Study Participant Daily Surveys, Support Person, Daily Surveys and Passive Monitoring.
Time Frame: Baseline until study completion (approximately 12 weeks)
Population: ASD and Typically Developing Population. The number analyzed includes participants who were evaluable at each timepoint.
Measure: Number; unit: Participants
Groups:
- Typically Developing Adults: Participants will be 18-45 years old, with IQ scores of 70 or above
- Typically Developing Adolescents: Participants will be 13-17 years old, with IQ scores of 70 or above
- Typically Developing Children: Participants will be 5-12 years old, with IQ scores of 70 or above
Arm/Group | Low-Functioning ASD Adults | High-Functioning ASD Adults | Typically Developing Adults | Low-Functioning ASD Adolescents | High-Functioning ASD Adolescents | Typically Developing Adolescents | Low-Functioning ASD Children | High-Functioning ASD Children | Typically Developing Children
Number analyzed (Participants) | 18 | 16 | 17 | 13 | 15 | 17 | 17 | 16 | 15
Participants
  Active Tests: number analyzed (Participants) | 18 | 16 | 17 | 13 | 11 | 17 | 17 | 10 | 15
  Active Tests | 10 | 12 | 13 | 7 | 11 | 6 | 6 | 10 | 8
  Conversation | 11 | 12 | 9 | 8 | 11 | 4 | 6 | 10 | 8
  Study Participant Daily Surveys | 11 | 11 | 13 | 4 | 9 | 6 | 6 | 7 | 8
  Support Person Daily Surveys | 14 | 12 | 13 | 9 | 11 | 6 | 6 | 12 | 8
  Passive Monitoring: number analyzed (Participants) | 5 | 13 | 17 | 8 | 8 | 17 | 5 | 5 | 15
  Passive Monitoring | 13 | 5 | 10 | 8 | 8 | 3 | 5 | 5 | 7

17. Secondary Outcome: Behaviour Rating Inventory of Executive Function for Children (BRIEF)
Description: The Behaviour Rating Inventory of Executive Function (BRIEF) parent questionnaire was designed to assess executive functioning of children with a wide spectrum of developmental and acquired neurological conditions, such as: Learning disabilities, Low birth weight, Attention-deficit/hyperactivity disorder, Tourette's disorder, Traumatic brain injury, Pervasive developmental disorders/autism (Gioia et al 2000).
  The pediatric Behavior Rating Inventory of Executive Function (BRIEF) consists of 86 caregiver reported items (three -point scale, N=never "1", S=sometimes "2", O= often "3" ) used to assess problems with executive functioning. The total score called global executive composite score which is calculated as the sum of the items and may range from 86 to 258 with higher total scores indicating more problems with executive functioning.
Time Frame: Baseline, Weeks 2 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | High-Functioning ASD Children | High-Functioning ASD Adolescents | Low-Functioning ASD Children | Low-Functioning ASD Adolescents
Number analyzed (Participants) | 16 | 15 | 17 | 13
Score on a Scale
  Baseline: number analyzed (Participants) | 16 | 15 | 17 | 12
  Baseline | 203.63 (27.95) | 189.50 (25.76) | 196.47 (31.97) | 184.08 (23.35)
  Week 2: number analyzed (Participants) | 16 | 13 | 14 | 11
  Week 2 | 197.13 (34.06) | 196.15 (24.32) | 194.36 (33.47) | 188.18 (29.17)
  Week 12: number analyzed (Participants) | 15 | 11 | 13 | 11
  Week 12 | 196.47 (35.84) | 190.82 (24.22) | 196.00 (31.28) | 189.55 (29.13)

18. Secondary Outcome: Behaviour Rating Inventory of Executive Function for Adults (BRIEF-A)
Description: The Behaviour Rating Inventory of Executive Function (BRIEF) parent questionnaire was designed to assess executive functioning of children with a wide spectrum of developmental and acquired neurological conditions, such as: Learning disabilities, Low birth weight, Attention-deficit/hyperactivity disorder, Tourette's disorder, Traumatic brain injury, Pervasive developmental disorders/autism (Gioia et al 2000).
  The adult Behavior Rating Inventory of Executive Function (BRIEF-A) consists of 75 caregiver reported items (three -point scale, N=never "1", S=sometimes "2", O= often "3") used to assess problems with executive functioning. The total score called global executive composite score which is calculated as the sum of the items and may range from 75 to 225 with higher total scores indicating more problems with executive functioning.
Time Frame: Baseline, Weeks 2 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | High-Functioning ASD Adults | Low-Functioning ASD Adults
Number analyzed (Participants) | 16 | 18
Score on a Scale
  Baseline: number analyzed (Participants) | 16 | 17
  Baseline | 150.06 (21.74) | 153.35 (25.61)
  Week 2: number analyzed (Participants) | 15 | 18
  Week 2 | 149.67 (22.64) | 156.83 (22.22)
  Week 12: number analyzed (Participants) | 14 | 18
  Week 12 | 152.43 (19.48) | 157.61 (24.48)

19. Secondary Outcome: Short Sensory Profile (SSP)
Description: The Short Sensory Profile (SSP) is a 38-item parent or caregiver reported questionnaire that probes for the effect of sensory processing anomalies on a person's ability to function in daily life. Item responses occur on a five-point Likert-rating scale from 1 (always occurs) to 5 (never occurs). The Short Sensory Profile was based on the Sensory Profile and provides 3 sets of standard scores depending on how the items are clustered: (1) domain scores, (2) factor scores and (3) a total score of all items. Total scores at the visits are reported.
  For the SSP, the possible total score can range between 38-190, with lower scores indicating more severe effect of sensory processing anomalies on a person's ability to function in daily life.
Time Frame: Baseline, Weeks 2 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a Scale
Groups:
- Low-Functioning (ASD Children: Participants will be 5-12 years old, with Intelligence Quotient (IQ) scores between 50-70
Arm/Group | High-Functioning ASD Children | High-Functioning ASD Adolescents | Low-Functioning (ASD Children | Low-Functioning ASD Adolescents
Number analyzed (Participants) | 16 | 15 | 17 | 13
Score on a Scale
  Baseline: number analyzed (Participants) | 16 | 14 | 16 | 13
  Baseline | 125.75 (23.76) | 132.86 (36.05) | 122.44 (26.84) | 138.73 (21.01)
  Week 2: number analyzed (Participants) | 16 | 13 | 14 | 10
  Week 2 | 128.19 (27.40) | 129.15 (37.99) | 127.07 (33.00) | 139.60 (22.44)
  Week 12: number analyzed (Participants) | 15 | 11 | 13 | 11
  Week 12 | 128.00 (25.99) | 136.91 (30.61) | 125.00 (25.14) | 136.73 (28.28)

20. Secondary Outcome: Vineland(TM)-II Survey
Description: The VinelandTM-II measures communication, daily living skills, socialization, motor skills (only in children up to 6 years) and maladaptive (not assessed in this study) behavior of individuals with developmental disabilities. The Survey Interview Form (i.e., semi -structured interview) will be administered to a participant's reliable caregiver in this study, during which the rater or clinician will ask to the caregiver open-ended questions relating to the participant's activities and behavior. Domain scores will be obtained for the individual domains of Socialization, Communication, Daily Living Skills, and motor skills (up to 6 years only) and used to calculate the VinelandTM-II Adaptive Behavior Composite score. Standardized scores on the adaptive behavior composite range from 20-160 with higher scores indicating better adaptive functioning. Values at visits are reported.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | High-Functioning ASD Children | High-Functioning ASD Adolescents | High-Functioning ASD Adults | Low-Functioning ASD Children | Low-Functioning ASD Adolescents | Low-Functioning ASD Adults
Number analyzed (Participants) | 16 | 15 | 16 | 17 | 13 | 18
Score on a Scale
  Baseline | 73.88 (8.08) | 75.07 (21.79) | 60.09 (23.71) | 69.41 (8.66) | 64.35 (6.33) | 44.86 (15.39)
  Week 12: number analyzed (Participants) | 13 | 13 | 14 | 17 | 13 | 17
  Week 12 | 72.08 (6.82) | 75.31 (13.65) | 59.86 (20.01) | 70.13 (9.00) | 63.23 (6.70) | 47.59 (15.28)

21. Secondary Outcome: Pediatric Quality of Life Inventory (PedsQL) Family Impact Scale
Description: The PedsQL™ Family Impact Module version 2 is a 36-item questionnaire which is completed by the caregiver and encompasses six scales covering 1) Physical Functioning (6 items), 2) Emotional Functioning (5 items), 3) Social Functioning (4 items), 4) Cognitive Functioning (5 items), 5) Communication (3 items), 6) Worry (5 items), and two scales measuring parent reported family functioning; 7) Daily Activities (3 items) and 8) Family Relationships (5 items). For each item a 5-point response scale is utilized (0=never a problem; 4=always a problem). Items are then reverse-scored and linearly transformed to a 0-100 scale (0-100, 1-75, 2-50, 3-25, 4-0), so that higher scores indicate better functioning (less negative impact). Scale Scores are computed as the sum of the items divided by the number of items answered (this accounts for missing data). If more than 50% of the items in the scale are missing, the Scale Score is not computed. Values at visits are reported.
Time Frame: Baseline, Weeks 2 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | High-Functioning ASD Children | High-Functioning ASD Adolescents | High-Functioning ASD Adults | Low-Functioning ASD Children | Low-Functioning ASD Adolescents | Low-Functioning ASD Adults
Number analyzed (Participants) | 16 | 15 | 16 | 17 | 13 | 18
Score on a Scale
  Baseline: number analyzed (Participants) | 16 | 14 | 15 | 17 | 12 | 17
  Baseline | 50.78 (15.21) | 52.58 (18.04) | 67.45 (15.47) | 54.13 (18.62) | 54.11 (15.10) | 63.44 (15.41)
  Week 2: number analyzed (Participants) | 16 | 13 | 15 | 14 | 11 | 18
  Week 2 | 52.60 (17.29) | 55.98 (23.13) | 65.23 (17.40) | 56.45 (20.05) | 53.47 (18.19) | 63.46 (18.63)
  Week 12: number analyzed (Participants) | 15 | 12 | 14 | 13 | 12 | 18
  Week 12 | 48.98 (19.36) | 59.95 (17.39) | 64.14 (17.80) | 57.43 (24.99) | 50.87 (16.99) | 60.65 (16.81)

22. Secondary Outcome: PedsQL Core Functioning Scale
Description: The PedsQL Cognitive Functioning Scale which contains six items will also be completed. The acute participant-completed forms (5 to 7 years, 8 to 12 years, 13 to 18 years, young adults, and adults) with a recall period of 7 days will be employed in this trial. For children aged 8 years and above, the PedsQL items are scored on a five-point Likert-type response scale (0=never a problem; 1=almost never a problem; 2=sometimes a problem; 3=often a problem; and 4=almost always a problem). For children age 5 to 7 years, scoring is based on a three point scale (0=Not at all, 2=Sometimes, 4=A lot). Items will be reverse-scored and linearly transformed to a 0-100 scale (0=100, 1=75, 2=50, 3=25, 4=0), so that higher scores indicate better health-related quality of life. For children aged 5-7 years, an administrator will read out the questions and the child will respond by pointing to one of three smiley faces. The values at visits are reported.
Time Frame: Baseline, Weeks 2 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a Scale
Groups:
- High-Functioning ASD Children-1: Participants will be 5-7 years old, with IQ scores of 70 or above
- High-Functioning ASD Children-2: Participants will be 8-12 years old, with IQ scores of 70 or above
- Low-Functioning ASD Children-1: Participants will be 5-7 years old, with Intelligence Quotient (IQ) scores between 50-70
- Low-Functioning ASD Children-2: Participants will be 8-12 years old, with Intelligence Quotient (IQ) scores between 50-70
Arm/Group | High-Functioning ASD Children-1 | High-Functioning ASD Children-2 | High-Functioning ASD Adolescents | High-Functioning ASD Adults | Low-Functioning ASD Children-1 | Low-Functioning ASD Children-2 | Low-Functioning ASD Adolescents | Low-Functioning ASD Adults
Number analyzed (Participants) | 4 | 12 | 15 | 11 | 5 | 12 | 13 | 11
Score on a Scale
  Baseline: number analyzed (Participants) | 4 | 12 | 15 | 6 | 5 | 9 | 9 | 7
  Baseline | 55.98 (4.82) | 64.22 (16.56) | 64.78 (16.63) | 61.78 (8.23) | 76.96 (21.17) | 62.44 (24.28) | 64.25 (22.33) | 56.83 (14.91)
  Week 2: number analyzed (Participants) | 4 | 12 | 13 | 6 | 4 | 9 | 8 | 7
  Week 2 | 46.74 (17.25) | 64.13 (20.15) | 73.66 (16.37) | 59.60 (10.04) | 71.20 (23.64) | 66.91 (15.50) | 57.74 (23.32) | 54.50 (11.23)
  Week 12: number analyzed (Participants) | 4 | 9 | 13 | 6 | 1 | 6 | 10 | 6
  Week 12 | 45.11 (22.20) | 70.53 (18.14) | 70.07 (14.96) | 59.60 (12.11) | 76.09 (0) | 66.30 (21.64) | 57.72 (22.83) | 56.70 (11.65)

23. Secondary Outcome: PedsQL Cognitive Functioning Scale
Description: as for outcome 22
Time Frame: Baseline, Week 2 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | High-Functioning ASD Children | High-Functioning ASD Adolescents | High-Functioning ASD Adults | Low-Functioning ASD Children | Low-Functioning ASD Adolescents | Low-Functioning ASD Adults
Number analyzed (Participants) | 16 | 15 | 16 | 17 | 13 | 18
Score on a Scale
  Baseline: number analyzed (Participants) | 16 | 15 | 16 | 17 | 12 | 17
  Baseline | 50.78 (15.21) | 52.58 (18.04) | 67.45 (15.47) | 54.13 (18.62) | 54.11 (15.10) | 63.44 (15.41)
  Week 2: number analyzed (Participants) | 16 | 13 | 15 | 14 | 11 | 18
  Week 2 | 52.60 (17.29) | 55.98 (23.13) | 65.23 (17.40) | 56.45 (20.05) | 53.47 (18.19) | 63.46 (18.63)
  Week 12: number analyzed (Participants) | 15 | 12 | 14 | 13 | 12 | 18
  Week 12 | 48.98 (19.36) | 59.95 (17.39) | 64.14 (17.80) | 57.43 (24.99) | 50.87 (16.99) | 60.65 (16.81)

ADVERSE EVENTS:
Time Frame: From baseline to the study completion- Week 12
Description: There was no Serious Adverse Events reported.
Groups:
- High-Functioning ASD Adolescent; High-Functioning ASD Adults; Low-Functioning ASD Adolescent; Low-Functioning ASD Adults; Healthy Control Adolescents: Participants will be 13-17 years old, with IQ scores of 70 or above
- Low-Functioning ASD Children; Healthy Control Children: Participants will be 5-12 years old, with IQ scores of 70 or above
- Healthy Control Adults: Participants will be 18-45 years old, with IQ scores of 70 or above
Arm/Group | High-Functioning ASD Children | High-Functioning ASD Adolescent | High-Functioning ASD Adults | Low-Functioning ASD Children | Low-Functioning ASD Adolescent | Low-Functioning ASD Adults | Healthy Control Children | Healthy Control Adolescents | Healthy Control Adults
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/15 | 0/16 | 0/17 | 0/13 | 0/18 | 0/15 | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/16 | 0/17 | 0/13 | 0/18 | 0/15 | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 1/16 | 0/15 | 0/16 | 0/17 | 0/13 | 0/18 | 1/15 | 0/15 | 0/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-Functioning ASD Children (N=16) | High-Functioning ASD Adolescent (N=15) | High-Functioning ASD Adults (N=16) | Low-Functioning ASD Children (N=17) | Low-Functioning ASD Adolescent (N=13) | Low-Functioning ASD Adults (N=18) | Healthy Control Children (N=15) | Healthy Control Adolescents (N=15) | Healthy Control Adults (N=17)
Medical Device Site Erythema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/75/NCT03611075/Prot_SAP_000.pdf